CLINICAL TRIAL: NCT05969236
Title: A Phase 1, First-in-Human, Single-center, Randomized, Double-masked, Placebo-controlled Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of MDI-1228_mesylate Ophthalmic Solution by Local Instillation in Adult Healthy Volunteers
Brief Title: A Study of MDI-1228_mesylate Ophthalmic Solution in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Medinno Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MDI-1228-I-AC
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Intervention Model Description: This study consists of two parts:
  * Part A: Single ascending dose in healthy volunteers
  * Part B: Multiple ascending doses in healthy volunteers
  The randomization code and the randomization list will be generated using SAS version 9.4 or the latest available version at time of randomization.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Including 2 single dose groups (Part A) and 2 multiple dose groups (Part B). Participants in experimental groups will receive MDI-1228_mesylate Ophthalmic Solution.
  Interventions: Drug: MDI-1228_mesylate Ophthalmic Solution
- Comparator Group (Placebo Comparator): One comparator group will be set for each of the 4 experimental groups, to a total of 4 comparator groups. Participants in comparator groups will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDI-1228_mesylate Ophthalmic Solution — MDI-1228_mesylate Ophthalmic Solution includes 2 strengths:
  * 0.1% (0.4 mL [0.4 mg] free base)
  * 0.3% (0.4 mL [1.2 mg] free base)
  Arms: Experimental Group
Drug: Placebo — The components employed in the placebo formulation are the same as those used for the active formulation except MDI-1228_mesylate is absent.
  Arms: Comparator Group

SUMMARY:
The main goal of this clinical trial is to evaluate the safety, tolerability and pharmacokinetics (PK) profiles* of MDI-1228_mesylate Ophthalmic Solution in healthy adult participants.

Participants will receive either of the following treatment:

* MDI-1228_mesylate Ophthalmic Solution, or
* Placebo**

Researchers will observe any changes in health (if any) in participants receiving the study treatment to evaluate the safety and tolerability*** of the study drug. Researchers will also collect several blood samples from participants to study PK profiles of the drug.

Note:

*PK profiles: how the drug interacts with the body. **placebo: a harmless substance that contains no active agents. ***tolerability: how well you can tolerate the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Weight ≥ 50 kg for males, ≥ 45 kg for females, with the BMI (BMI = weight[kg]/height[m]2) between 18 and 32 (inclusive) at screening.
2. The corrected visual acuity (CVA) of both eyes should be 6/6 or 20/20 (Snellen chart), with an intraocular pressure between 10 and 21 mmHg (inclusive) and a difference in intraocular pressure between the 2 eyes < 5 mmHg at screening.
3. Normal vital signs after ≥ 5 minutes resting supine or semi supine position:

   1. ≥ 90 mmHg and ≤160 mmHg (systolic blood pressure)
   2. ≥50 mmHg and ≤ 95 mmHg (diastolic blood pressure)
   3. ≥ 45 beats per minute (bpm) and ≤ 100 bpm (heart rate)
   4. Body temperature ≥35.5℃ and ≤37.7℃
   5. Respiratory Rate≥12 breaths/minute and≤22 breaths/minute
4. Standard 12-lead ECG parameters after ≥5 minutes resting in supine or semi-supine position with PR ≥ 120 ms and ≤ 220 ms, QRSD < 120 ms, QTcF ≤ 450 ms for males and ≤ 470 ms for females, and otherwise normal ECG (all data limits are based on average readings of the ECGs) at screening.
5. Females must be non-pregnant and non-lactating, and either surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy), or use highly effective contraceptive method as assessed by the PI (OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD) from screening until study completion, including the follow up period for at least 30 days after the last dose of study drug, or be post-menopausal for ≥ 12 months. Post-menopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels at screening for amenorrheic female participants. Females who are abstinent from heterosexual intercourse as part of their usual lifestyle will also be eligible for participation.
6. Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and admission and be willing to have additional pregnancy tests as required throughout the study.
7. Males must be surgically sterile (> 30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, the participant and his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective contraceptive method as assessed by the PI from screening until study completion, including the follow up period, for at least 30 days after the last dose of study drug. Acceptable methods of contraception include the use of condoms and the use of an effective contraceptive for the female partner (WOCBP) that includes: OCPs, long- acting implantable hormones, injectable hormones, a vaginal ring, or an IUD. Male participants whose female partner is post-menopausal, and participants who are abstinent from heterosexual intercourse as part of their usual lifestyle and are not planning to conceive will also be eligible.
8. Male participants must agree to refrain from donating sperm and female participants from donating ova from screening until study completion, including the follow up period, for at least 90 days after the last dose of study drug.
9. Provides written informed consent and is willing and able to undergo all study procedures and attend the scheduled follow up visit/s per protocol.
10. Are willing to consume clinical research unit (CRU) provided meals.
11. Have no neck or back issues which prevents the participant having their head tilted back for dosing at the discretion of the Investigator.
12. Males and females aged 18 to 55 years old (inclusive)
13. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, safety laboratory tests, and ECG. A potential participant with a clinical abnormality or laboratory parameters outside the normal reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. The Investigator may discuss with the local MM and Sponsor MM as required.
14. Have no abnormal results or abnormal not clinically significant (as determined by the Investigator) results of ocular examinations of both eyes (including slit-lamp examination, corneal fluorescein staining test, light response pupil test, extraocular movement test, dilated fundus examination)

Exclusion Criteria:

1. Have a current or past history of clinically significant circulatory system diseases, respiratory disorders, hepatobiliary disorders, digestive disorders, urinary system diseases, renal disorders, endocrine disorders, immune system disorders, malignancies, metabolic disorders, mental disorders, or nervous system diseases that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk to the participant by virtue of their participation in the study. Participant with a history of uncomplicated kidney stones (defined as spontaneous passage and no recurrence in the last 5 years); uncomplicated cholecystectomy; Gilbert's syndrome; a past history of being treated by non-current depression may be enrolled in the study at the discretion of the Investigator. Participants with a history of childhood asthma (without hospitalization) that has symptomatically resolved and remains untreated may participant.
2. Have healed eye disorders (such as infection, trauma) in either eye within 1 month prior to the first dose.
3. Have a history of intraocular surgery and laser eye surgery in either eye.
4. Used any ocular products (including various eye drops or eye gel) within 14 days or 5 half-lives (whichever is longer) prior to screening.
5. Wore contact lenses within 2 days prior to baseline (Day -1) or need to wear contact lenses throughout the clinical study.
6. Current evidence or history of COVID-19 or influenza-like illness as defined by fever (> 37.7°C) and 2 or more of the following symptoms within 7 days before dosing: cough, sore throat, runny nose, sneezing, limb/joint pain, headache, vomiting/diarrhea in the absence of a known cause, other than influenza or COVID-19 infection.
7. A positive pre-study HIV, Hepatitis B surface antigen or positive Hepatitis C antibody result at screening.
8. Participants who are intolerant of venipuncture blood collection or have poor venous access and/or have a history of fear of needles and hemophobia.
9. Used Janus kinase (JAK) inhibitors or immunosuppressants or any other prescription drugs, traditional Chinese medicines or Chinese patent medicines within 4 weeks prior to Day -1; or used over-the-counter (OTC) drugs or health products within 2 weeks prior to Day -1, unless with a washout period of more than 5 half-lives for products with a longer half-life. The Principal Investigator may review medication on a case-by-case basis to determine if its use would compromise participant safety or interfere with study procedures or data interpretation.
10. Was vaccinated within 2 weeks prior to screening or plan to be vaccinated during the study.
11. Had major surgery within 6 months prior to screening or plan to undergo surgery during the study.
12. Participants who smoked more than 5 cigarettes/pipes/vaping per day on average or excessive use of any nicotine product (> 5 products on average per day) within 3 months prior to screening and not able to abstain from smoking from screening to end of study (EoS).
13. Any other serious medical condition or abnormality that, in the Investigator's judgment, precludes the participant's safe participation in and completion of the study.
14. A positive pre-study drug or alcohol screen. A positive drug or alcohol screen test result may be verified by re-testing (up to 1 false positive result permitted) and may be followed up at the discretion of the Investigator.
15. History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of > 21 units for males or > 14 units for females. One unit is equivalent to 10 g of alcohol and the following can be used as a guide: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (30 mL) measure of spirits.
16. The participant is unwilling to abstain from alcohol consumption from 24 hours prior to dosing until discharge from the CRU, and for 24 hours prior to all other outpatient visits to the CRU.
17. Known history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric, human or humanized antibodies, fusion proteins, MDI-1228_mesylate Ophthalmic Solution excipients, any material used for assessments (e.g., fluorescein, tropicamide, etc), or a history of drug or other allergy including severe allergic reaction that in the opinion of the Investigator contraindicates their participation.
18. Participation in a clinical trial within 30 days before randomization; use of any experimental therapy within 30 days or 5 half-lives prior to randomization, whichever is greater; or use of any biologic therapy within 12 weeks or 5 half-lives prior to randomization, whichever is greater.
19. Pregnant or breastfeeding WOCBP.
20. Donation within the last 3 months of > 499 mL whole blood or within 2 weeks of any volume of plasma.
21. Participant unable to provide written informed consent or participant under guardianship.
22. Unwilling or unable to follow protocol requirements, including attendance at follow up visit/s.
23. Any history of severe ocular trauma in either eye at any time.
24. Any history of any refractive surgery procedure within the past 6 months of the screening visit in either eye.
25. Current or chronic history of clinically significant ocular disease within the past 3 months of screening visit in either eye.
26. Current or chronic history of ocular infection (bacterial, viral, or fungal) or corneal irritation within the past 3 months of screening visit in either eye.
27. Abnormal tearing, OR expected regular use of prescription or expected use of OTC tear substitutes within 4 weeks prior to Day -1, and for the duration of the study.
28. Previous or expected use of ocular (topical, periocular, intravitreal), local (inhaled or nasal), or systemic steroid or glucocorticoid medications within 4 weeks prior to Day -1, and for the duration of the study.
29. At the Investigator's or delegate's discretion, any participants who have a history of any significant ocular conditions in either eye that would contraindicate the use of the study medication, or that might affect the study conduct, or the interpretation of the study results.
30. Clinically significant findings as determined by the Investigator in other ocular examinations (e.g., conjunctival hyperemia grade >1, corneal fluorescein staining score ≥ 2, or other chronic or acute eye disorders).
31. History of clinically significant ocular disease (glaucoma, retinal detachment, iritis, uveitis, herpetic keratitis, etc.) that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk to the participant by virtue of their participation in the study.
32. Presence of an ocular pathology such as blepharitis, conjunctivitis, uveitis, or any other ocular infection or inflammation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Part A and B - Incidence and severity of all systemic or ocular treatment emergent adverse events (TEAEs) | From first dose to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Systemic or ocular TEAEs will be collected from spontaneous reports and direct observation.
  The investigator will make an assessment of intensity for each TEAE and assign it to one of the Common Terminology Criteria for Adverse Events (CTCAE) categories: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (life-threatening), and grade 5 (death).
Part A and B - Assessment of vital sign measurement results - respiratory rate | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Respiratory rate (breaths/minute) will be measured while the participant is at rest in a supine or semi-supine position (after ≥ 5 minutes resting supine or semi-supine), to monitor and record any abnormal clinically significant changes from baseline and incidence of such changes after treatment until the last visit.
Part A and B - Assessment of vital sign measurement results - heart rate | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Heart rate (beats/minute) will be measured while the participant is at rest in a supine or semi-supine position (after ≥ 5 minutes resting supine or semi-supine), to monitor and record any abnormal clinically significant changes from baseline and incidence of such changes after treatment until the last visit.
Part A and B - Assessment of vital sign measurement results - blood pressure | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Blood pressure (mmHg) will be measured while the participant is at rest in a supine or semi-supine position (after ≥ 5 minutes resting supine or semi-supine), to monitor and record any abnormal clinically significant changes from baseline and incidence of such changes after treatment until the last visit.
Part A and B - Assessment of vital sign measurement results - body temperature | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Body temperature (℃) will be measured while the participant is at rest in a supine or semi-supine position (after ≥ 5 minutes resting supine or semi-supine), to monitor and record any abnormal clinically significant changes from baseline and incidence of such changes after treatment until the last visit.
Part A and B - Assessment of physical examination results - general appearance | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of general appearance (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - head, eyes, ears, nose, and throat (HEENT) | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of HEENT (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - neck (including thyroid and nodes) | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of neck (including thyroid and nodes) (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - cardiovascular system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of cardiovascular system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - respiratory system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of respiratory system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - gastrointestinal system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of gastrointestinal system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - renal system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of renal system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - neurological system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of neurological system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - musculoskeletal system | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of musculoskeletal system (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of physical examination results - skin | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Assessment of skin (normal/abnormal) will be performed at screening, and may be performed at various scheduled/unscheduled time points if deemed necessary by the Investigator, to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of 12-lead electrocardiogram (ECG) results - heart rate | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  12-lead ECG measurements will be performed to monitor and record any abnormal clinically significant changes in heart rate (beats/min) as well as the result interpretation from baseline and incidence of such changes after treatment until the last visit. All ECG measurements will be recorded in triplicate (repeat for 3 times), with 1- to 2-minute intervals between ECG readings.
Part A and B - Assessment of 12-lead ECG results - PR interval | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  12-lead ECG measurements will be performed to monitor and record any abnormal clinically significant changes in PR interval (milliseconds) as well as the result interpretation from baseline and incidence of such changes after treatment until the last visit. All ECG measurements will be recorded in triplicate, with 1- to 2-minute intervals between ECG readings.
Part A and B - Assessment of 12-lead ECG results - QRSD interval | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  12-lead ECG measurements will be performed to monitor and record any abnormal clinically significant changes in QRSD interval (milliseconds) as well as the result interpretation from baseline and incidence of such changes after treatment until the last visit. All ECG measurements will be recorded in triplicate, with 1- to 2-minute intervals between ECG readings.
Part A and B - Assessment of 12-lead ECG results - QT interval corrected with Fridericia Formula (QTcF) | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  12-lead ECG measurements will be performed to monitor and record any abnormal clinically significant changes in QTcF (milliseconds) as well as the result interpretation from baseline and incidence of such changes after treatment until the last visit. All ECG measurements will be recorded in triplicate, with 1- to 2-minute intervals between ECG readings.
Part A and B - Assessment of 12-lead ECG results - RR interval | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  12-lead ECG measurements will be performed to monitor and record any abnormal clinically significant changes in RR interval (milliseconds) as well as the result interpretation from baseline and incidence of such changes after treatment until the last visit. All ECG measurements will be recorded in triplicate, with 1- to 2-minute intervals between ECG readings.
Part A and B - Ophthalmic assessment - corrected visual acuity (CVA) | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  CVA (measured using Snellen chart) will be assessed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - intraocular pressure | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Intraocular pressure (mmHg) will be assessed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - light response pupil test | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Light response pupil test (positive/negative) will be performed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - extraocular movement test | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Extraocular movement test will be performed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - slit-lamp examination | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Slit-lamp examination will be performed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - corneal fluorescein staining test | From screening to end of study (EOS, Day 7±1 day in Part A, Day 14±1 day in Part B)
  Corneal fluorescein staining test will be performed to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Ophthalmic assessment - dilated fundus examination | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Dilated fundus examination will be performed at screening, Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes from baseline and the incidence of such changes after treatment until the last visit.
Part A and B - Assessment of hematology results - red blood cell distribution width | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in red blood cell distribution width (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - hemoglobin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in hemoglobin (g/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - hematocrit | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in hematocrit (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - red blood cell count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in red blood cell count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - white blood cell count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in white blood cell count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - absolute neutrophil count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in absolute neutrophil count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - neutrophil percentage | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in neutrophil percentage (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - absolute lymphocyte count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in absolute lymphocyte count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - lymphocyte percentage | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in lymphocyte percentage (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - absolute monocyte count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in absolute monocyte count (cells/μL)) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - monocyte percentage | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in monocyte percentage (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - absolute basophil count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in absolute basophil count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - basophil percentage | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in basophil percentage (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - absolute eosinophil count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in absolute eosinophil count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - eosinophil percentage | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in eosinophil percentage (%) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - platelet count | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in platelet count (cells/μL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - mean cell hemoglobin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in mean cell hemoglobin (pg/cell) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - mean cell volume | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in mean cell volume (fL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - mean cell hemoglobin concentration | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in mean cell hemoglobin concentration (g/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of hematology results - mean platelet volume | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Hematology tests will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in mean platelet volume (fL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of coagulation results - international normalized ratio (INR) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  A coagulation test will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in INR from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of coagulation results - activated partial thromboplastin time (aPTT) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  A coagulation test will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in aPTT (seconds) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of coagulation results - prothrombin time (PT) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  A coagulation test will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in PT (seconds) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - sodium | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood sodium (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - potassium | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood potassium (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - chloride | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood chloride (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - calcium | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood calcium (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - bicarbonate | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes from baseline in blood bicarbonate (mmol/L) and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - albumin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes from baseline in blood albumin (g/dL) and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - total protein | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in total protein (g/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - creatinine | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood creatinine (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - creatine kinase | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood creatine kinase (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - estimated glomerular filtration rate (GFR) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes from baseline in estimated GFR (mL/min) and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - urea | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood urea (μmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - aspartate aminotransferase (AST) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in AST (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - alanine aminotransferase (ALT) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in ALT (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - gamma glutamyl transpeptidase (GGT) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in GGT (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - alkaline phosphatase (ALP) | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in ALP (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - phosphate | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood phosphate (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - total bilirubin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in total bilirubin (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - direct bilirubin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in direct bilirubin (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - indirect bilirubin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in indirect bilirubin (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - amylase | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood amylase (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - cholesterol | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in cholesterol (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - high density lipoprotein (HDL)/cholesterol ratio | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in HDL/cholesterol ratio from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - high density lipoprotein (HDL) cholesterol | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in HDL cholesterol (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - low density lipoprotein (LDL) cholesterol/high density lipoprotein (HDL) cholesterol ratio | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in LDL/HDL cholesterol ratio from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - low density lipoprotein (LDL) cholesterol | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in LDL cholesterol (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - non-high density lipoprotein (HDL) cholesterol | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in non-HDL cholesterol (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - triglycerides | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in triglycerides (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - uric acid | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in uric acid (μmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - lactate dehydrogenase | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in lactate dehydrogenase (units/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - magnesium | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood magnesium (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - glucose | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in blood glucose (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - anion gap | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in anion gap (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - adjusted calcium | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in adjusted calcium (mmol/L) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of blood biochemistry results - globulin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Blood biochemistry will be measured at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in globulin (g/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - pH | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in pH from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - specific gravity | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in specific gravity from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine glucose | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine glucose (negative/+/++/+++) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine protein | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine protein (negative/+/++/+++) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine bilirubin | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine bilirubin (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine ketones | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine ketones (negative/+/++/+++) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine blood | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine blood (negative/+/++/+++) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine nitrite | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine nitrite (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - urine urobilinogen | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in urine urobilinogen (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of urinalysis results - leucocyte esterase | From screening to end of treatment (Day 2 in Part A, Day 8 in Part B)
  Urinalysis will be performed at screening, baseline (not required if screening assessment done within 3 days), Day 2 visit (Part A) or Day 8 visit (Part B) to monitor and record any abnormal clinically significant changes in leucocyte esterase (mg/dL) from baseline and the incidence of such changes after treatment until last visit.
Part A and B - Assessment of scores of conjunctival hyperemia | From pre-dose to post-dose (Day 2 in Part A, Day 8 in Part B)
  Scores of conjunctival hyperemia (0 to 4 scores, a higher score indicates a more severe condition) will be assessed to record the change from the pre-dose (Day -1) scores to the post-dose scores (Day 2 for Part A, Day 8 for Part B) in the study eye.
Part A and B - Assessment of scores of corneal staining | From pre-dose to post-dose (Day 2 in Part A, Day 8 in Part B)
  Scores of corneal staining (0 to 5 scores, a higher score indicates a more severe condition) will be assessed to record the change from the pre-dose (Day -1) scores to the post-dose scores (Day 2 for Part A, Day 8 for Part B) in the study eye.

SECONDARY OUTCOMES:
Part A - Maximum concentration (Cmax) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  Cmax means the highest concentration a drug reaches in the plasma after administration. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A and B - Time to maximum concentration (Tmax) of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day in Part A, Day 14±1 day in Part B)
  Tmax refers to the time a drug takes to reach the highest concentration in the plasma after administration. It will be measured after the subject receives a single dose (Part A) or multiple doses (Part B) of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A and B - Half-life (T1/2) of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day in Part A, Day 14±1 day in Part B)
  T1/2 refers to the time a drug takes to be eliminated to half of the highest concentration in the plasma after administration. It will be measured after the subject receives a single dose (Part A) or multiple doses (Part B) of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A - Systemic clearance (CL or CL/F) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  Systemic CL refers to the total volume of fluid cleared of drug from the body per unit of time, usually expressed in mL/min. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A - Volume of distribution (Vd) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  Vd refers to fluid volume that would be required to contain the amount of drug present in the body at the same concentration as in the plasma. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A - Mean retention time (MRT) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  MRT reflects the average time a drug molecule spends in the body. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A - Area under curve until time t (AUC0-t) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  AUC0-t refers to area under the plasma concentration-time curve until time t and reflects the actual body exposure to drug after administration at time t. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part A - Area under curve until infinity (AUC0-∞) of MDI-1228_mesylate Ophthalmic Solution after a single dose of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 7±1 day)
  AUC0-∞ refers to area under the plasma concentration-time curve until infinity and reflects the total body exposure to drug. It will be measured after the subject receives a single dose of MDI-1228_mesylate Ophthalmic Solution by instillation into the study eye (2 drops).
Part B - Trough concentration at steady state (Css_min) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  Css_min means the lowest concentration of drug in the blood within a steady-state dosing interval. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).
Part B - Maximum plasma concentration at steady state (Css_max) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  Css_max means the highest concentration of drug in the blood observed after intermittent dosage administration. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).
Part B - Average plasma concentration at steady state (Css_av) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  Css_av means the average drug concentration reached during a steady-state intermittent dosing interval. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).
Part B - Clearance (CL or CL/F) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  CL means the volume of fluid cleared of drug from the body per unit of time, usually expressed in mL/min. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).
Part B - Area under the plasma concentration-time curve at steady state (AUCss) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  AUCss reflects the exposure of drug in the body at steady state. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).
Part B - Coefficient of fluctuation (DF) of MDI-1228_mesylate Ophthalmic Solution following multiple doses of MDI-1228_mesylate Ophthalmic Solution | Post-first dose on Day 1 to EOS (Day 14±1 day)
  DF reflects difference between the highest and lowest concentration of drug in the body at steady state. It will be measured after administration of multiple doses of MDI-1228_mesylate Ophthalmic Solution by conjunctival instillation (2 drops).

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, PhD, Principal Investigator — CMAX Clinical Research; Liang Lu, PhD, Study Director — Shanghai Medinno Pharmaceutical Technology Co., Ltd.
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No